CLINICAL TRIAL: NCT01024972
Title: Dantrolene in the Prevention and Treatment of Cerebral Vasospasm in Subarachnoid Hemorrhage
Brief Title: Safety Study of Dantrolene in Subarachnoid Hemorrhage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-13441
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Dantrolene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dantrolene (Experimental): Dantrolene 1.25mg/kg IV every 6 hours x 7 days
  Interventions: Drug: Dantrolene
- Placebo (Placebo Comparator): Equiosmolar volume (5% Mannitol)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dantrolene — Dantrolene 1.25mg/kg IV (includes 5% mannitol) every 6 hours x 7 days
  Other Names: Dantrium
  Arms: Dantrolene
Drug: Placebo — equiosmolar volume (5% mannitol) every 6 hours x 7 days
  Other Names: Free water/5% mannitol solution
  Arms: Placebo

SUMMARY:
Subarachnoid hemorrhage (SAH) is a devastating acute brain injury due to bleeding onto the brain surface from a ruptured aneurysm. Cerebral vasospasm (cVSP; critical narrowing of brain arteries) is a known complication after SAH and significantly increases disability and death after SAH. Vasospasm is difficult to treat and can lead to stroke. Animal studies have shown that the muscles in the artery wall play a role in cVSP.

Dantrolene has been FDA approved and extensively used in clinical practice as a muscle relaxant for more than 30 years. It has been shown to provide some benefit in animal studies of cVSP, as well as in a small number of humans. However, the first human studies have only been observational and over a short period of time.

This study will evaluate the safety and tolerability of intravenous dantrolene given every 6 hours over seven days to patients with or at risk for cVSP after SAH. The goal is to determine if future efficacy studies should be done to determine if treatment with Dantrolene may improve the outcome of patients with cVSP after SAH.

DETAILED DESCRIPTION:
Once eligibility criteria are met, patients will be randomized to either dantrolene-IV or placebo (equiosmolar, volume-equivalent sterile water with 5% mannitol as dantrolene-IV also contains 5% mannitol). Study subjects will be visited daily by a study nurse to determine side effects, tolerability, record hemodynamic measures and laboratory values. Patients will have daily serum Na, osmolality, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALK) measured. In addition, daily bedside transcranial doppler will be performed by a blinded examiner. Patients will undergo cerebral angiograms per clinical routine. Angiographic measurements of arterial narrowing will be performed by a blinded radiologist. Specific stop criteria are pre-defined.

ELIGIBILITY:
Inclusion Criteria:

* Documented aneurysmal SAH by computed tomography angiography (CTA), magnetic resonance angiography (MRA) or angiography
* Secured aneurysm (coiled or clipped)
* Enrollment achievable within 14 days after SAH

Exclusion Criteria:

* Pregnancy
* Prior history of cirrhosis or hepatitis B/C, or any two of the following three liver enzymes elevated to greater than: ALT >120 Units/L, AST >120 Units/L, alkaline phosphatase >345 Units/L (three times upper limit of normal)
* Patients on verapamil
* Patients with brain edema and/or elevated intracranial pressure (>25mm Hg)
* Patients treated with hypertonic saline or mannitol prior to enrollment
* Patients with too severe SAH with low likelihood of survival (Hunt & Hess 5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Muehlschlegel, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMASS Medical School / UMass Memorial Medical Center, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Salomone S, Soydan G, Moskowitz MA, Sims JR. Inhibition of cerebral vasoconstriction by dantrolene and nimodipine. Neurocrit Care. 2009;10(1):93-102. doi: 10.1007/s12028-008-9153-0. Epub 2008 Oct 16. PMID 18923817
- [Background] Muehlschlegel S, Rordorf G, Bodock M, Sims JR. Dantrolene mediates vasorelaxation in cerebral vasoconstriction: a case series. Neurocrit Care. 2009;10(1):116-21. doi: 10.1007/s12028-008-9132-5. Epub 2008 Aug 12. PMID 18696267
- [Background] Muehlschlegel S, Sims JR. Dantrolene: mechanisms of neuroprotection and possible clinical applications in the neurointensive care unit. Neurocrit Care. 2009;10(1):103-15. doi: 10.1007/s12028-008-9133-4. Epub 2008 Aug 12. PMID 18696266
- [Background] Muehlschlegel S, Rordorf G, Sims J. Effects of a single dose of dantrolene in patients with cerebral vasospasm after subarachnoid hemorrhage: a prospective pilot study. Stroke. 2011 May;42(5):1301-6. doi: 10.1161/STROKEAHA.110.603159. Epub 2011 Mar 31. PMID 21454813
- [Result] Muehlschlegel S, Carandang R, Hall W, Kini N, Izzy S, Garland B, Ouillette C, van der Bom IM, Flood TF, Gounis MJ, Weaver JP, Barton B, Wakhloo AK. Dantrolene for cerebral vasospasm after subarachnoid haemorrhage: a randomised double blind placebo-controlled safety trial. J Neurol Neurosurg Psychiatry. 2015 Sep;86(9):1029-35. doi: 10.1136/jnnp-2014-308778. Epub 2014 Oct 24. PMID 25344064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with aSAH were screened for eligibility between 10/2009 and 10/2012. Inclusion criteria were aSAH ≥18 years, aneurysm fully secured by coiling or clipping, Hunt&Hess grade <5, modified Fisher Scale >1, ALT, AST, AlkPhos <3x upper limit of normal, serum Na (sNa) ≥135mmol/L and no mannitol or hypertonic saline prior to drug infusion.
Pre-assignment Details: Routine patient management: All aSAH patients were treated according to our institutional protocol following published aSAH critical care guidelines, including admission to our closed neuroscience intensive care unit (neuroICU) with board-certified neurointensivist as the primary attending.
Groups:
- Dantrolene: Dantrolene 1.25mg/kg IV every 6 hours x 7 days
  Dantrolene vs. Placebo: Dantrolene 1.25mg/kg IV (includes 5% mannitol) or equiosmolar placebo (5% mannitol) every 6 hours x 7 days
- Placebo: Equiosmolar volume (5% Mannitol)
  Dantrolene vs. Placebo: Dantrolene 1.25mg/kg IV (includes 5% mannitol) or equiosmolar placebo (5% mannitol) every 6 hours x 7 days
Period: Overall Study
Arm/Group | Dantrolene | Placebo
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dantrolene: Intravenous Datrolene 1.25 mg/kg (includes 5% mannitol) every 6 hours for seven days.
- Placebo: Equiosmolar volume (5% mannitol) every 6 hours for seven days.
- Total: Total of all reporting groups
Arm/Group | Dantrolene | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12) | 52 (11) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15 | 9 | 24
  Hispanic/Latino | 0 | 6 | 6
  African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hyponatremia
Description: Number of subjects who developed hyponatremia (sNa ≤132mmol/L)
Time Frame: Seven days
Measure: Number; unit: participants
Groups:
- Placebo: equiosmolar, volume-equivalent sterile water with 5% mannitol every 6 hours x 7 days.
Arm/Group | Dantrolene | Placebo
Number analyzed (Participants) | 16 | 15
participants | 7 | 10

2. Secondary Outcome: Liver Toxicity
Description: Number of subjects who developed liver toxicity as evidenced by Liver Function Test elevation greater than 5 times the upper limit of normal.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Dantrolene | Placebo
Number analyzed (Participants) | 16 | 15
participants | 1 | 0

3. Secondary Outcome: In-hospital Mortality
Description: Number of subjects who expired during hospitalization.
Time Frame: up to 90 days
Measure: Number; unit: participants
Arm/Group | Dantrolene | Placebo
Number analyzed (Participants) | 16 | 15
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Dantrolene | Placebo
Serious Adverse Events (participants affected / at risk) | 4/16 | 2/15
Other Adverse Events (participants affected / at risk) | 12/16 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dantrolene (N=16) | Placebo (N=15)
Neurological deterioration (Nervous system disorders) | 2 (2) | 1 (1) — Neurological deterioration requiring osmotherapy
Liver toxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) — Liver function test elevation greater than 5 times upper limit of normal
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Drug administration error (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dantrolene (N=16) | Placebo (N=15)
Venous infiltration (Vascular disorders) | 4 (4) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Non-(ST wave)-elevation myocardial infarction
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Placebo group consisted of free water with 5% mannitol to achieve the same equiosmolar solution as IV-D which requires reconstitution in free water. Unable to differentiate whether hyponatremia or brain oedema was due to IV-D or its solution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No